CLINICAL TRIAL: NCT00737971
Title: A Randomized, Parallel Group, Masked Clinical Study to Evaluate the Efficacy of Triamcinolone and Bevacizumab Through Intravitreal Injection With Individual or Simultaneous Drugs to Treatment of Diabetic Macular Edema
Brief Title: Efficacy Study of Triamcinolone and Bevacizumab Intravitreal for Treatment of Diabetic Macular Edema
Acronym: ATEMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rubens Belfort Jr. (Other)
Responsible Party: Sponsor-Investigator, Rubens Belfort Jr., Head Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108/08
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Macular Edema
Keywords: avastin; bevacizumab; triamcinolone; diabetic macular edema; macular edema; intravitreal injection
MeSH Terms: conditions — Macular Edema | interventions — Bevacizumab; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Avastin intravitreal injection D0, Week 4, Week 8
  Interventions: Drug: Bevacizumab intravitreal
- B (Active Comparator): Triamcinolone intravitreal injection
  Interventions: Drug: Triamcinolone
- C (Active Comparator): Avastin + Triamcinolone intravitreal injection simultaneously
  Interventions: Drug: Triamcinolone + Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab intravitreal — Bevacizumab intravitreal 0.05 ml/1.25 mg - administered on D0, Week 4, Week 8
  Other Names: Avastin
  Arms: A
Drug: Triamcinolone — Intravitreal 0.1 ml/4 mg, D0, Week 4 and Week 8
  Arms: B
Drug: Triamcinolone + Bevacizumab — Intravitreal triamcinolone 0.1 ml/4 mg + bevacizumab 0.05 ml/1.25 mg simultaneously on D0, week 4, Week 8
  Other Names: triamcinolone + avastin
  Arms: C

SUMMARY:
Triamcinolone and Bevacizumab Intravitreal for Treatment of Diabetic Macular Edema

DETAILED DESCRIPTION:
Efficacy Study of Triamcinolone and Bevacizumab Intravitreal for Treatment of Diabetic Macular Edema

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at least
* Diagnosis of diabetes mellitus (type 1 or type 2. any one of the following will be considered to be sufficient evidence that diabetes is present:

  * current regular use of insulin for the treatment of diabetes
  * current regular use of oral hypoglycemic agents for the treatment of diabetes
  * diabetes as defined by american Diabetes Association (ADA)
  * symptoms of diabetes (polyuria, polydipsia, and unexplained weight loss) or eighth-hour fasting plasma glucose > 126 mg/dl
* Diabetic macular edema clinically observable associated with diabetic retinopathy:

  * without prior foveal treatment with laser therapy
  * if photocoagulation or peripherical or macular laser, at least 3 months
  * absence of macular ischemia by fluorescein angiography on baseline visit
* BCVA score between 20 letters (20/400 ETDRS)e 70 letters (20/40 ETDRS) in the study eye measured by the ETDRS method at qualification/baseline visit
* Retinal thickness > 275um by OCT
* One eye per patient will be chosen for the study. In case of both eye eligible, it will be chosen an eye to be treated with study medication and another eye treated with laser
* Taught hyaloid syndrome

Exclusion Criteria:

* Uncontrolled systemic disease
* Initiation of medical therapy for diabetes or a change from oral hypoglycemic agents to insulin therapy within 4 months prior to the qualification visit
* Renal failure requiring hemodialysis or peritoneal dialysis within 6 months prior to the qualification visit
* Any ocular condition in the study eye that in the opinion of the investigator would prevent a 2 lines improvement of visual acuity (e.g. severe macular ischemia)
* Presence of branch retinal vein occlusion, central retinal vein occlusion, uveitis, pseudophakic cystoid edema or any other condition in the study eye which could be contributing to macular edema
* Presence of an epiretinal membrane in the study eye
* History of IOP elevation in response to steroid treatment in either eye
* History of glaucoma or optic nerve head change consistent with glaucoma damage
* Ocular hypertension requiring more than 1 anti-glaucoma medication to maintain IOP < 11mmhg at qualification visit
* Presence of anterior chamber intraocular lens in the study eye
* Active optic disc or retinal neovascularization in the study eye at qualification visit
* Active or history of choroidal neovascularization in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measurement of visual acuity (E Snellen) | monthly

SECONDARY OUTCOMES:
Tonometry | monthly
Measurement of retinal thickness by OCT | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, Principal Investigator — Federal University of São Paulo / Dept. of OPhthalmology
Locations (1):
- Federal University of Sao Paulo - Dept. of Ophthalmology / Vision Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
data presented in several congresses: ARVO 2010-- poster ARVO 2011, WOC BERLIN 2010, WOC ABU DABHI 2012 (partial data) CBO 2014 (final data)